CLINICAL TRIAL: NCT04738409
Title: Ovarian Hyperandrogenism in Adolescent Girls and Concomitant Metabolic Changes, Oxidative Stress, Inflammation, Oral Health and Their Relation to Diet
Brief Title: Ovarian Hyperandrogenism in Normal and Excessive Body Weight Adolescent Girls and Their Relation to Diet (HAstudy)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Poznan University of Physical Education (Other)
Collaborators: National Science Centre, Poland (Other Government); Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Małgorzata Mizgier, Assistant Professor, Poznan University of Physical Education
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HA000001
Record Dates: First submitted 2021-01-21; First posted 2021-02-04 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ov/Ob group (Experimental): PCOS subjects (Overweight/Obesity)
  Interventions: Other: Lifestyle intervention; Other: Effects of AIDiet intervention to improve diet quality, immuno-metabolic health in normal and overweight PCOS girls
- N group (Experimental): PCOS subjects (Normal weight)
  Interventions: Other: Lifestyle intervention; Other: Effects of AIDiet intervention to improve diet quality, immuno-metabolic health in normal and overweight PCOS girls
- H group (No Intervention): Healthy control subjects

INTERVENTIONS:
Other: Lifestyle intervention — The purpose of the research is to evaluate the potential of a multidimensional lifestyle program for PCOS girls. The primary aim is to verify the effectiveness of a 16-week AID intervention vs. HCD (combined with PA&T), in terms of improvement in androgens level and immune-metabolic risk parameters
  Arms: N group; Ov/Ob group
Other: Effects of AIDiet intervention to improve diet quality, immuno-metabolic health in normal and overweight PCOS girls — The purpose of the intervention is to evaluate the effectiveness of the anti-inflammatory diet (AIDiet) among normal weight (N) and overweight/obese (Ov/Ob) women with PCOS.
  Arms: N group; Ov/Ob group

SUMMARY:
The objective was

1. to check whether serum androgen levels and concomitant metabolic changes, oxidative stress and inflammation in adolescent girls with hyperandrogenism may be related to diet.
2. to identify the factors that increase the risk of being overweight and of obesity among adolescents with clinical features of PCOS, related to diet and DEA (Disordered Eating Attitudes)
3. to investigate the relationships between markers of oxidation and markers of Systemic Inflammation and macronutrients intake
4. to assess the relation between oral health of girls with PCOS (including condition of periodontium and dental caries) and their dietary habits, hormonal, metabolic and oxidative and inflammatory status.

DETAILED DESCRIPTION:
Hyperandrogenism in women is a state of increased androgen production, manifested by irregular menstrual cycles, a more frequent incidence of infertility, metabolic syndrome, oxidative stress, and inflammation, as well as acne and hirsutism. In addition to ovulation disorders and the multifollicular ovaries structure in an ultrasound examination, hyperandrogenism is a typical clinical feature of the Polycystic Ovary Syndrome (PCOS), which is diagnosed in approximately 8.6% of adolescent girls. Excessive body weight makes it difficult to diagnose at an early stage of the disease and intensifies metabolic and hormonal disorders, as well as those related to oxidative stress and inflammation of the body. Some research studies suggest that PCOS may negatively affect oral health of women, increasing the risk of periodontal problems.

The main purpose of this research was to check whether serum androgen levels and concomitant metabolic changes, oxidative stress and inflammation in adolescent girls with hyperandrogenism may be related to diet.

The investigators aimed to identify the factors that increase the risk of being overweight and of obesity among adolescents with clinical features of PCOS, related to diet and DEA(Disordered Eating Attitudes).

The objective was also to investigate the relationships between markers of oxidation and markers of Systemic Inflammation and macronutrients intake, such as carbohydrates and fiber, protein (animal, plant), fats and cholesterol in normal and overweight/obese girls with clinical features of PCOS.

Additionally, the investigators would like to evaluate the relation between oral health of girls with PCOS (including condition of periodontium and dental caries) and their dietary habits, hormonal, metabolic and oxidative and inflammatory status.

ELIGIBILITY:
Inclusion Criteria:

The criteria for the patient's inclusion were based on the 2003 Rotterdam criteria, with the presence of at least two of the following:

* written consent for inclusion (girls and their parents)
* clinical and/or biochemical hyperandrogenism (hirsutism with moderate to severe acne, and/or elevation of serum total testosterone or free testosterone,
* oligoovulation (based on oligomenorrhea defined as bleeding episodes occurring less than 8 times per year or secondary amenorrhea),
* polycystic ovarian picture in an ultrasound examination (at least 12 follicles in each ovary each measuring 2-9 mm in diameter and/or ovarian volume >10 mL).

Exclusion Criteria:

* any systemic disease, thyroid dysfunction, diabetes, congenital adrenal hyperplasia, Cushing syndrome, hyperprolactinemia suggestive of pituitary adenoma and androgen-secreting tumors
* medications of continuous use,
* the use of hormonal therapy or antibiotics in the past three months,
* vitamin or supplements use,
* alcohol consumption
* smoking

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood parameters | 2018-2022
  Hormonal and biochemical parameters, including follicle-stimulating hormone (FSH), luteinizing hormone (LH), total testosterone, androstenedione, estradiol, dehydroepiandrosterone (DHEA-S), Sex Hormone Binding Globulin (SHBG), fasting glucose and fasting insulin, total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C), and triglycerides (TG), 17 OH-Progesterone, Prolactin, Cortisol, Thyroid-stimulating hormone (TSH), will be measured in the morning after overnight fasting.
Anthropometric Assessment | 2018-2022
  Body mass index BMI: derived from measured body height (m) and body weight (kg) as body weight / height². Weight will be measured to the nearest 0.1 kg using digital medical scales. Height will be measured with a stadiometer attached to the scales.
  Waist circumference (WC) will be measured to the nearest 0.1 mm using anthropometric tape between the lower border of rib margin and the upper border of iliac crest (WC-mid).
Body Composition | 2018-2022
  Body composition will be assessed with a body composition analyzer (BIA method). The measurements of fat mass (FM) will be expressed as a percentage (%) and kilograms (kg).

OTHER OUTCOMES:
Disordered Eating Attitudes | 2018-2022
  Eating behavior will be assessed with a standard Eating Attitudes Test-26 (EAT-26), a self-administrated questionnaire.
Inflammation and Oxidative Stress | 2018-2022
  Serum concentrations of the inflammation markers: Interleukin 1 (IL-1), Interleukin 6 (IL-1), Tumor Necrosis Factor (TNF-α), C-reactive protein (CRP) and the markers of oxidation: malondialdehyde, total antioxidant capacity will be measured with a commercial ELISA assay kits
Nutrition evaluation | 2018-2022
  Nutrition evaluation will be conducted by continuous recording of all consumed foodstuffs, dishes and beverages, specifying home measures and weight (3-day food record method and food frequency method FFQ). Data will be analysed using The Aliant computer program (Cambridge Diagnostics).
Oral Health Assessment | 2018-2022
  * Severity of gingivitis expressed as a Gingival Index (GI)
  * Presence of gingivitis assessed based on the percentage of sites bleeding upon probing BOP%.
  * The subgingival microflora assessed on the basis of the number of specific bacteria isolated from gingival sulci of every individual and the percentage of patients affected by specific periodontal pathogens.
  * Salivary levels of TNF-alfa, IL-6, IL-1B, uric acid used to assess and compare the inflammation in oral environment.
  * Testosteron in saliva used to compare androgenic status of patients with PCOS and healthy controls.
Evaluation of physical activity | 2018-2022
  International Physical Activity Questionnaire will be applied, including records of the type and specific character of the training and activity, its duration, intensity and frequency.
The Data From The Child's Health Book | 2018-2022
  Collected from the child's health book regarding newborn body weight and term of delivery. The incidence of macrosomia (body weight over 4000 g) or low birth weight, LBW (body weight less than 2500 g) was assessed on the basis of the newborn's body weight. The full term of delivery (term births) will be assessed for deliveries that occur between 38-42 weeks of pregnancy, while preterm births will be defined as those deliveries between 23 weeks and 37 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata Mizgier, PhD, Principal Investigator — Poznan University of Phisical Education, Dietetic Department; Justyna Opydo-Szymaczek, PhD, Principal Investigator — Poznan University of Medical Scienses; Grażyna Jarząbek-Bielecka, PhD, Principal Investigator — Poznan University of Medical Scienses
Locations (2):
- Poland (2):
  - Poznan University of Medical Sciences, Poznan
  - Poznan University of Physical Education, Poznan

REFERENCES:
- [Derived] Mizgier M, Wieckowska B, Formanowicz D, Lombardi G, Brozek A, Nowicki M, Durkalec-Michalski K, Kedzia W, Jarzabek-Bielecka G. Effects of AIDiet intervention to improve diet quality, immuno-metabolic health in normal and overweight PCOS girls: a pilot study. Sci Rep. 2024 Feb 12;14(1):3525. doi: 10.1038/s41598-024-54100-1. PMID 38347150
- [Derived] Mizgier M, Watrowski R, Opydo-Szymaczek J, Jodlowska-Siewert E, Lombardi G, Kedzia W, Jarzabek-Bielecka G. Association of Macronutrients Composition, Physical Activity and Serum Androgen Concentration in Young Women with Polycystic Ovary Syndrome. Nutrients. 2021 Dec 24;14(1):73. doi: 10.3390/nu14010073. PMID 35010948
- [Derived] Mizgier M, Jarzabek-Bielecka G, Formanowicz D, Jodlowska-Siewert E, Mruczyk K, Cisek-Wozniak A, Kedzia W, Opydo-Szymaczek J. Dietary and Physical Activity Habits in Adolescent Girls with Polycystic Ovary Syndrome (PCOS)-HAstudy. J Clin Med. 2021 Aug 5;10(16):3469. doi: 10.3390/jcm10163469. PMID 34441766
- [Derived] Mizgier M, Jarzabek-Bielecka G, Wendland N, Jodlowska-Siewert E, Nowicki M, Brozek A, Kedzia W, Formanowicz D, Opydo-Szymaczek J. Relation between Inflammation, Oxidative Stress, and Macronutrient Intakes in Normal and Excessive Body Weight Adolescent Girls with Clinical Features of Polycystic Ovary Syndrome. Nutrients. 2021 Mar 10;13(3):896. doi: 10.3390/nu13030896. PMID 33801995

DOCUMENTS (1):
  • Study Protocol (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT04738409/Prot_000.pdf